CLINICAL TRIAL: NCT04951960
Title: The Impact of Higher Positive End Expiratory Pressure on Patient-Ventilator Asynchrony in Patients With Acute Respiratory Distress Syndrome: a Cross-Over Randomized Trial
Brief Title: The Impact of Higher Positive End Expiratory Pressure on Patient-Ventilator Asynchrony
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Osaka University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PEEPPVA
Record Dates: First submitted 2020-11-01; First posted 2021-07-07 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2020-11

CONDITIONS: Critical Illness
Keywords: patient ventilator asynchrony; positive end expiratory pressure
MeSH Terms: conditions — Critical Illness; Patient-Ventilator Asynchrony

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants, their legal representatives, and outcomes assessor are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group from higher PEEP to lower PEEP (Other): Patient allocated for this arm are received from higher to lower PEEP setting.
  Interventions: Other: Higher PEEP setting; Other: Lower PEEP setting
- A group from lower PEEP to higher PEEP (Other): Patient allocated for this arm are received from lower to higher PEEP setting.
  Interventions: Other: Higher PEEP setting; Other: Lower PEEP setting

INTERVENTIONS:
Other: Higher PEEP setting — PEEP levels are determined according to the higher PEEP-FiO2 tables set plateau pressure less than 30 cmH2O. The duration of measurement at each PEEP levels is 1 hour.
Other: Lower PEEP setting — PEEP levels are determined according to the lower PEEP-FiO2 tables set plateau pressure less than 30 cmH2O. The duration of measurement at each PEEP levels is 1 hour.

SUMMARY:
Patient-ventilator asynchrony is known to frequently occur during lung protective ventilation in patients with ARDS. Previous clinical studies showed that patient-ventilator asynchrony was associated with worse outcome in ICU. Therefore, strategies to reduce patient-ventilator asynchrony need to be established promptly. Several asynchronies, e.g., breath stacking are caused by vigorous spontaneous breathing effort. Recently, the investigators' group found that higher positive end expiratory pressure (PEEP) reduced the intensity of spontaneous breathing effort of in severe ARDS model (rabbits, pigs) and patients with ARDS. Thus, the investigators conjectured that higher PEEP may reduce the intensity of spontaneous breathing effort and thereby reduce patient-ventilator asynchrony during protective ventilation strategy, compared with lower PEEP in patients with ARDS.

DETAILED DESCRIPTION:
The cross-over study will enroll 10 participants fulfilled with the criteria of Berlin definition of moderate-to-severe ARDS and under mechanical ventilation in intensive care unit (ICU) at Osaka University Hospital. Informed consent will be obtained by legal representatives. After obtaining informed consent, participants will be randomly assigned to one of two groups: "higher PEEP - lower PEEP" or "lower PEEP - higher PEEP". PEEP, either higher or lower, will be set according to higher or lower PEEP/FIO2 table. The depth of sedation will be monitored quantitively and maintained to be the same throughout the protocol. The intensity of spontaneous breathing activity will be assessed with esophageal balloon manometry and electrical activity of diaphragm. At each PEEP setting, asynchrony index will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≧ 18 years old
2. Patients with moderate to severe ARDS under mechanical ventilation＊ ＊ Definition of moderate to severe ARDS is as per the Berlin definition (PaO2/FiO2 ≦ 200 mmHg with PEEP ≧ 5 cmH2O)

Exclusion Criteria:

1. Lack of informed consent
2. Continuous neuromuscular blockade at enrollment
3. DNR (do-not-resuscitate)
4. Moribund patient not expected to survive 24 hours
5. Massive hemoptysis
6. Increased intracranial pressure (> 18 mmHg)
7. Existence or high risk of pneumothorax
8. Known pregnancy
9. Actual body weight exceeding 1 kg/cm
10. Patient judged to be inappropriate for the trial by intensivist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Asynchrony index of all types of patient ventilator asynchrony at higher and lower PEEP. | Through study completion (up to 24 hours)

SECONDARY OUTCOMES:
Asynchrony index of each types of patient ventilator asynchrony at higher and lower PEEP. | Through study completion (up to 24 hours)
The intensity of spontaneous breathing effort measured by esophageal manometry at higher and lower PEEP | Through study completion (up to 24 hours)
Minute volume at higher and lower PEEP | Through study completion (up to 24 hours)
The efficiency of diaphragmatic contraction measured by electrical activity of diaphragm at higher and lower PEEP. | Through study completion (up to 24 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Yoshida, M.D., Ph.D., Principal Investigator — Osaka University
Locations (1):
- Osaka University Hospital, Suita, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No